CLINICAL TRIAL: NCT05055050
Title: A Window of Opportunity Phase I Study of UGN-201 in Patients With Bladder Cancer Undergoing Radical Cystectomy
Brief Title: A Window of Opportunity Phase I Study of UGN-201 in Patients With Bladder Cancer Undergoing Radical Cystectomy Protocol #: 2021-0630
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Interim Analysis
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0630; NCI-2021-09539 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-09-07; First posted 2021-09-23 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer; Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UGN-201 Pre Radical Cystectomy (Experimental): UGN-201 200 mg/50ml
  Interventions: Drug: UGN-201

INTERVENTIONS:
Drug: UGN-201 — Intravesical 200 mg /50 ml x 1 dose
  Other Names: imiquimod intravesical solution

SUMMARY:
he primary objective is to characterize the safety profile of UGN-201 in patients with urothelial carcinoma undergoing radical cystectomy.

Corresponding primary endpoint: Toxicity of concern (TOX) will be monitored until 30 days after surgery or until the patient meets the surgery prevention or delay TOX definition below, whichever comes first. A patient will be considered to have a TOX if any of the following apply:

* Any 30-day grade 3 or higher surgical complication at least possibly related to UGI-201
* Any toxicity at least possibly related to the treatment that prevents surgery or delays it more than 12 weeks from date of cystectomy decision with MDACC Urologist. Missing/delayed surgery due to progression or withdrawal not related to toxicity will not count as a TOX event. Rapid progression is not seen with UGN-201. For such a patient, TOX monitoring will follow for 30 days after the administered dose of UGN-201.
* Death between the start of study and the 30-day post-surgical assessment will count if it is toxic death at least possibly related to the UGN-201 or surgery. Deaths clearly unrelated to treatment will not count as an event.

Adverse events will be recorded using CTCAE v5 and surgical complications will be recorded using Clavien-Dindo classification.

Exploratory objectives are:

* To evaluate the efficacy of UGN-201 by pathologic T0 and ≤ pT1 rate (pathologic down-staging) after neoadjuvant treatment with UGN-201, in patients with NMBIC and MIBC undergoing radical cystectomy, respectively.
* To assess the immunological/biomarker changes in tumor tissues, peripheral blood, and urine in response to UGN-201 treatment in patients with bladder cancer undergoing radical cystectomy and to explore any potential association between these biomarker measures and antitumor activity.

Patients with MIBC will be defined as having a response if their pathologic stage is pT1 stage or less. Patients with NMIBC will be defined as having a response if their pathologic stage is pT0.

Immunologic and other biomarker measures will be recorded by laboratory standards for each measure.

DETAILED DESCRIPTION:
Primary Objective:

-To characterize the safety profile of UGN-201 in patients with urothelial carcinoma undergoing radical cystectomy.

Exploratory Objectives:

* To evaluate the efficacy of UGN-201 by pathologic T0 and ≤ pT1 rate (pathologic downstaging) after neoadjuvant treatment with UGN-201, in patients with NMBIC and MIBC undergoing radical cystectomy, respectively.
* To assess the immunological/biomarker changes in tumor tissues, peripheral blood, stool and urine in response to UGN-201 treatment in patients with bladder cancer undergoing radical cystectomy and to explore any potential association between these biomarker measures and antitumor activity.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible for participation in this trial, the subject must:

* Be willing and able to provide written informed consent
* Be ≥ 18 years of age
* Have histological confirmation of predominant urothelial cancer (either non-muscle invasive or muscle invasive). Patients whose tumors are found to be invasive should not have stage 3 or greater disease.
* Have absence of metastatic disease as determined by conventional imaging studies and be considered a good surgical candidate by the treating physician.
* Be willing to participate in the collection of blood, tissue, stool, and urine for banking and future correlative studies as specified in the Study Flow Chart (Section 6.0).
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days of treatment initiation.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 30 days after the last dose of study medication.

  10. Male subjects of childbearing potential (Section 5.7.2) must agree to use an adequate method of contraception as outlined in Section 5.7.2- Contraception, starting with the first dose of study therapy through 30 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

-Patients must consent to the MD Anderson Immunotherapy Platform laboratory protocol PA13-0291.

Exclusion Criteria

The subject must be excluded from participating in the trial if the subject:

* Is currently participating and receiving UGN-201 or has participated in a study of an investigational agent and received UGN-201 or used an investigational device within 4 weeks of the first dose of study treatment.
* Has ≥ cT3 and/or cN+ and/or cM+ urothelial carcinoma of the bladder, non-predominant urothelial carcinoma or histologic variants, such as small cell, carcinosarcoma, squamous cell or adenocarcinoma.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a known history of hypersensitivity to UGN-201 or any of its excipients.
* Has had prior systemic anti-cancer therapy for the treatment of bladder cancer. Prior intravesical therapies, whether BCG, chemotherapy or otherwise, will remain eligible Has cT3 or bulkier urothelial carcinoma of the bladder
* Has any other malignancy diagnosed within 2 years of screening with the exception of basal or squamous cell skin cancer, or non-invasive cancer of the cervix, or any other cancer deemed by the treating physician to be of low risk for progression or patient morbidity during the study period.
* Has known metastatic disease as determined by conventional staging studies.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has a clinically significant active infection requiring systemic therapy and cannot be resolved prior to initiating treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating physician.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Clinically significant urethral stricture that would preclude passage of a urethral catheter.
* History of pelvic radiotherapy.
* History of neurogenic bladder.
* History of active urinary retention.
* History of any other condition that would prohibit normal voiding.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a vaccine within 30 days of initiation of study therapy. Exceptions will be made for inactivated seasonal influenza and COVID-19 vaccines at the discretion of the treating physician. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed under any circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To establish the safety profile of UGN-201 in patients with urothelial carcinoma undergoing radical cystectomy. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Neema Navai, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org